CLINICAL TRIAL: NCT05074212
Title: Aesthetic Outcome of Complex Linear Closure vs Second Intention Healing for Cutaneous Surgical Procedures Performed Below the Knee: a Randomized, Blind Control Trial
Brief Title: Aesthetic Outcome of Complex Linear Closure vs Second Intention Healing: Below the Knee
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 1515109
Record Dates: First submitted 2021-09-29; First posted 2021-10-12 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-05

CONDITIONS: Wound Heal; Wound of Skin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Complex Linear Closure (Experimental): The study participant will receive two layers of sutures to close the wound.
  Interventions: Other: Factorial Assignment
- Second Intention Healing (Experimental): The study participant will not have any sutures placed.
  Interventions: Other: Factorial Assignment

INTERVENTIONS:
Other: Factorial Assignment — At the follow-up visit, two blinded observers will record their scores independently using the physician observer scar assessment score instrument (POSAS).

SUMMARY:
The purpose of this study is to determine whether complex linear closure vs second intention healing for cutaneous wounds below the knee affects esthetic outcomes (primary outcome). As secondary outcome, the study team plans to look at patient quality of life measures and complications. This will be a prospective, 2-arm, randomized, evaluator-blinded clinical trial. One half of the patients will receive repair by complex linear closure and the other half of the patients will undergo second intention healing. Three-months post-surgery, the scar will be evaluated via the patient observer scar assessment scale (POSAS), a validated scar instrument, as well as the trace-to-tape method, an objective outcome measure for linear postoperative scars. In addition, patients will be provided a validated quality of life survey to complete. Any adverse events will also be recorded.

DETAILED DESCRIPTION:
When a cutaneous wound is created following Mohs micrographic surgery and standard excisions, a decision is made to either allow the wound to heal by second intention ("leave open") or repair the wound ("close"). The decision may depend on patient characteristics, wound location, wound size or wound characteristics.

When the decision is made to repair the wound, the majority of wounds are reconstructed using two layers of sutures: a deep (subcutaneous) layer and a top (cutaneous) layer.

This study aims to investigate whether complex linear closure versus second intention healing for cutaneous surgical procedures performed below the knee affects wound cosmesis. In other words, the study team would like to determine which of the following yields a more cosmetically appealing scar: below the knee wound that is closed in a linear fashion or below the knee wound that is left open to heal on its own. The study team also plans to look at quality of life measures via validated surveys and complications.

Randomized control trials comparing these two methods appear to be lacking. A randomized trial looked at second intention healing vs primary simple closure following 4mm or 8mm punch biopsies on the arm, back or thigh1. Besides this study, no other information could be found in the literature on randomized trials comparing linear closure vs second intent for cutaneous wounds below the knee. The study team hopes that this study will provide new insight in cutaneous surgery.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Able to give informed consent themselves
* Patient scheduled for cutaneous surgical procedure below the knee with a lesion excision diameter of at least 1 cm.
* Willing to return for follow up visit

Exclusion Criteria:

* Incarceration
* Under 18 years of age
* Pregnant Women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 172 (Estimated)
Dates: Start 2022-01-10 (Actual); Primary Completion 2030-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
POSAS | 3-12 months
  The primary outcome is the sum of the average components of the Observer portion of the Patient and Observer Scar Assessment Scale (POSAS). The observer scale of the POSAS consists of six items (vascularity, pigmentation, thickness, relief, pliability and surface area).
  All items are scored on a scale ranging from 1 ('like normal skin') to 10 ('worst scar imaginable'). The sum of the six items results in a total score of the POSAS observer scale. Categories boxes are added for each item. Furthermore, an overall opinion is scored on a scale ranging from 1 to 10.
Mean Scar Width | 3-12 months
  Mean scar width will be measured using the trace-to-tape method.

SECONDARY OUTCOMES:
Occurrence of Complications | 3-12 months
  Occurrence of any complications from the treatment including: spitting sutures, dehiscence, infection, necrosis, bleeding, and hematoma.
Quality of Life Measures (DLQI) | 3-12 months
  The DLQI aim is to measure how much patient's skin problem has affected their life.The DLQI consists of 10 questions concerning patients' perception of the impact of skin diseases on different aspects of their health-related quality of life over the last week.

CONTACTS AND LOCATIONS:
Locations (1):
- University of California, Davis, Department of Dermatology, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: No